CLINICAL TRIAL: NCT02552979
Title: Atopy Patch Test in Children With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: Si524/2011
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Atopic Dermatitis; Food Allergy
Keywords: atopic dermatitis; atopic patch test
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: atopic patch test

SUMMARY:
Positive reactions in atopy patch test in children with atopic dermatitis.

DETAILED DESCRIPTION:
The prevalence of food allergy seems to be increasing, which might explain the increased demand for reliable evaluation of patients with suspected food-related gastrointestinal symptoms. Little is known about the diagnostic accuracy of atopy patch tests(APT) in the clinical practice. APT seems to have a better specificity than the IgE methods and seems to reflect late-phase clinical reactions.The aims of this study were to evaluate:

(i) The prevalence of positive reaction of APTs for atopic dermatitis (ii)Positive reaction of APT compare with skin prick test. (iii)Positive reaction of APT using lyophilized food vs commercially available food extracts. (iv)Side effect or adverse

ELIGIBILITY:
Inclusion Criteria:

* Patients who had history of atopic dermatitis

Exclusion Criteria:

* Who have dermographism
* Who have chronic disease eg. autoimmune disease, immune deficiency, cancer or allergic disease
* Pregnant women
* Who receive antihistamine, topical steroid and systemic steroid > 20 mg/day within 7 days prior study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
atopic patch test in atopic dermatitis children | 1 year